CLINICAL TRIAL: NCT01911286
Title: Comparison of Two Strategies to Realize Apnea Test for the Diagnostic of Brain in Potentiel Organ Donors.
Acronym: APNEE REA
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: APNEE REA
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Alternative Method of Apnea Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- Standard group: Apnea test according to the recommendation
  Interventions: Procedure: Apnea test - Standard
- CPAP group: Apnea test with CPAP connection
  Interventions: Procedure: Apnea test - CPAP

INTERVENTIONS:
Procedure: Apnea test - Standard
  Groups: Standard group
Procedure: Apnea test - CPAP
  Groups: CPAP group

SUMMARY:
Clinical diagnostic of brain death requires a non-reactive coma, absence of brain stem reflex, and absence of spontaneous breathing. The confirmation of absence of spontaneous breathing is established the apnea test (according to the American Academy of Neurology's Guidelines). However this test may lead to complications (acute hypoxemia, ventilatory and cardiocirculatory disorders) and reduces significantly the number of lung transplants. Some data suggest modifying the apnea test : replace the ventilator switching off with continuous positive airway pressure (CPAP) use. These studies showed that this alternative method (CPAP) increased the level of lung harvest but they were not sufficient because these studies were monocentric with little patients,. That why the aim of the present study is to compare the standard strategy and CPAP strategy with a prospective, multicenter,cluster trial; each center will use the method of apnea test which it uses usually.

ELIGIBILITY:
Inclusion Criteria:

* Age : from 18 to 75 years
* Neurological signs evoking cerebral ischemia

Exclusion Criteria:

* Severe hypoxemia (PaO2/FiO2 < 200) with controlled ventilation (FiO2: 100%)
* Hypothermia < 36°C
* Obesity (BMI ≥ 40) with documented hypopnoea
* Intractable hypotension despite optimal filling and catecholamine doses > 1µg.Kg.min
* Patients with contraindication for organs harvesting.
* Documented chronic respiratory failure
* Progressive infectious acute respiratory disease
* Family opposition to subject's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentiel organs donors in brain death.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Eligibility to lung harvest | 2 years

SECONDARY OUTCOMES:
Levels of hypoxemia | 2 years
Arterial blood gas after apnea test | 2 years
Rate of ventilatory impairment | 2 years
Rate of cardiocirculatory impairment | 2 years
Rate of apnea test interruption | 2 years
Number of lung transplantation realization | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michel PINSARD, Hospital Practitioner, Principal Investigator — Poitiers University Hospital
Locations (17):
- France (17):
  - Angers University Hospital, Angers
  - Angoulême Hospital, Angoulême
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Tours University Hospital, Chambray-lès-Tours
  - Sud Francilien Hospital, Corbeil-Essonnes
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - La Rochelle Hospital, La Rochelle
  - Limoges University Hospital, Limoges
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - Orléans Hospital, Orléans
  - Cochin University Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University hospital, Rennes
  - Saintes Hospital, Saintes
  - Toulon University Hospital, Toulon